CLINICAL TRIAL: NCT05229406
Title: Healthy Minds Program (HMP) App Dosage Study
Brief Title: Healthy Minds Program App Dosage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1578; MSN227550 (Other Grant/Funding Number: UW Madison); 2019-1578 (Other: UW Madison); A171600 (Other: UW Madison); EDUC/COUNSELING PSYCH (Other: UW Madison); 01/21/2022 (Other: UW Madison); 1K23AT010879-01 (NIH)
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Depression; Anxiety; Psychological Distress
Keywords: depression; anxiety; behavioral symptoms
MeSH Terms: conditions — Depression; Anxiety Disorders; Behavioral Symptoms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to two groups in a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-minute app usage (Experimental): Participants will be asked to use the HMP app for 5-minutes per day.
  Interventions: Behavioral: HMP app
- 15-minute app usage (Experimental): Participants will be asked to use the HMP app for 15-minutes per day.
  Interventions: Behavioral: HMP app

INTERVENTIONS:
Behavioral: HMP app — The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose.

SUMMARY:
The study will evaluate the effectiveness of the Healthy Minds Program (HMP) meditation app on participants experiencing depression and/or anxiety. Participants will be assigned to use the HMP app 5- or 15-minutes per day for 4 weeks.

DETAILED DESCRIPTION:
Depression and anxiety are highly common, but access to evidence-based treatments is limited. Meditation training delivered through mobile health (mHealth) technology may increase access to effective strategies. However, the necessary dosage of meditation practice to produce benefits is unknown. This project will investigate the feasibility, acceptability, and preliminary effectiveness of the HMP app for depression and/or anxiety and the feasibility of randomly assigning participants to practice dosages. Further, the project will provide a preliminary evaluation of the linkages between practice dosage and outcomes assessed retrospectively and in-the-moment via ecological momentary assessment (EMA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Access to a smartphone or device capable of downloading HMP app
* Self-reported willingness to complete 1-2 min survey 4 times per day on phone for 4 weeks
* Able to speak, read, and write in English
* PROMIS Depression or PROMIS Anxiety >55

Exclusion Criteria:

* Meditation retreat experience
* Regular meditation practice (weekly practice for over 1 year OR daily practice within the previous 6 months)
* Previous practice under the instruction of a meditation teacher, other than in the context of an introductory course
* PROMIS Depression >70
* AUDIT C score greater than or equal to 4 for men, and greater than or equal to 3 for non-men (any other genders)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be de-identified and listed in public data registries (e.g., OSF) based on the publication of preregistered study hypotheses on a manuscript by manuscript basis.
Time Frame: Data may be shared following analysis and publication or upon request.
Access Criteria: Researcher consent. Any reasonable request will be granted.

REFERENCES:
- [Derived] Dyer RL, Zimmerman KM, Zhao X, Xie Q, Dahl CJ, Quanbeck A, Goldberg SB. Developing meditation practice in individuals with elevated psychological distress via a meditation app intervention: An implementation science-informed qualitative investigation of barriers and facilitators. Psychol Serv. 2025 Jul 10:10.1037/ser0000980. doi: 10.1037/ser0000980. Online ahead of print. PMID 40638276
- [Derived] Xie Q, Dyer RL, Lam SU, Frye C, Dahl CJ, Quanbeck A, Nahum-Shani I, Davidson RJ, Goldberg SB. Understanding the Implementation of Informal Meditation Practice in a Smartphone-Based Intervention: A Qualitative Analysis. Mindfulness (N Y). 2024 Feb;15(2):479-490. doi: 10.1007/s12671-024-02304-x. Epub 2024 Jan 22. PMID 39070019

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from February 2022 to June 2022.
Period: Overall Study
Arm/Group | 5-minute App Usage | 15-minute App Usage
Started | 46 | 46
Completed | 45 | 44
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- 5-minute App Usage: Participants will be asked to use the HMP app for 5-minutes per day.
  The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose.
- 15-minute App Usage: Participants will be asked to use the HMP app for 15-minutes per day.
  The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose.
- Total: Total of all reporting groups
Arm/Group | 5-minute App Usage | 15-minute App Usage | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.72 (11.48) | 31.85 (14.68) | 31.28 (13.12)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 41 | 34 | 75
  Male | 5 | 8 | 13
  Other Gender | 0 | 4 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic White | 5 | 3 | 8
  American Indian | 1 | 1 | 2
  Asian | 9 | 9 | 18
  Black | 1 | 2 | 3
  Multiracial | 1 | 3 | 4
  White | 29 | 27 | 56
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 46 | 92

OUTCOME MEASURES:

1. Primary Outcome: Randomization Rate: Number of Participants Who Were Randomized and Completed EMA Assessments and Activities in the HMP App
Description: Percentage of those randomized completing ecological momentary assessment (EMA) assessments and activities in the Healthy Minds Program (HMP) app
Time Frame: Baseline to post-test (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
Participants | 46 | 46

2. Primary Outcome: Dosage Adherence: Number of Participants Adhering to Their Dosage Greater Than or Equal to 50 Percent of the Days
Description: Number of participants adhering to their assigned dosage greater than or equal to 50 percent of the days. This was assessed directly through the HMP app.
Time Frame: Baseline to post-test (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
Participants | 22 | 16

3. Primary Outcome: Percentage of EMA Completed
Description: Percentage of EMA assessments that were completed
Time Frame: Baseline to post-test (week 4)
Measure: Mean (Standard Deviation); unit: percentage of EMA assessments complete
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
percentage of EMA assessments complete | 82.71 (32.82) | 78.61 (41.00)

4. Primary Outcome: Study Completion Rate
Description: Percentage of participants completing pre- and post-test measures
Time Frame: Baseline to post-test (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
Participants | 45 | 44

5. Primary Outcome: Number of Participants Completing Practices ≥50% of Days
Description: Number of participants completing practices ≥50% of days
Time Frame: Baseline to post-test (week 4)
Measure: Count of Participants; unit: Participants
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
Participants | 32 | 26

6. Primary Outcome: Modified System Usability Scale (MSUS)
Description: The MSUS is a 10-item questionnaire where participants report their experience of the usability of a product, in this case the HMP app. It is scored on a 1- to 5-point Likert scale where 1 = strongly disagree and 5 = strongly agree. The result was rescaled to range from 0 to 100 with higher scores indicate higher usability.
Time Frame: Post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 45 | 44
score on a scale | 84.56 (10.86) | 83.66 (14.21)

7. Primary Outcome: Change in Attitudes Towards Psychological Online Interventions (ATPOI)
Description: The ATPOI is a 16-item questionnaire where participants report their perception of psychological online interventions. It is scored on a 1- to 5-point Likert scale where 1 = totally disagree and 5 = totally agree. Mean scores are reported for a total possible range of scores is 1 to 5 where higher scores indicate more positive attitudes towards psychological online interventions.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 3.30 (0.39) | 3.20 (0.36)
  T2 Post-Test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-Test Week 4 | 3.45 (0.50) | 3.47 (0.64)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.15 (0.47) | 0.27 (0.44)

8. Primary Outcome: HMP App Utilization: Minutes
Description: Minutes of meditation practice completed
Time Frame: Baseline to post-test (week 4)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
minutes | 100.85 (66.13) | 201.76 (144.61)

9. Primary Outcome: HMP App Utilization: Days
Description: Number of days the app was accessed.
Time Frame: Baseline to post-test (week 4)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
days | 17.28 (7.00) | 14.72 (7.89)

10. Primary Outcome: HMP App Utilization: Number of Activities
Time Frame: Baseline to post-test (week 4)
Measure: Mean (Standard Deviation); unit: activities
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
activities | 57.65 (32.40) | 51.43 (44.91)

11. Secondary Outcome: Change in Composite of Patient-Reported Outcomes Measurement Information System (PROMIS) Depression and PROMIS Anxiety
Description: Psychological distress will be computed as a composite of the PROMIS Depression and PROMIS Anxiety measures. We will use the computer adaptive version of both measures which have a mean of 50 and a standard deviation of 10. A composite will be computed by average across T-scores. T-scores range from 10 to 90 with higher scores indicating higher depression or anxiety.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
T-score
  T1 baseline | 60.93 (5.38) | 61.08 (5.24)
  T2 post-test (week 4): number analyzed (Participants) | 45 | 44
  T2 post-test (week 4) | 57.28 (5.63) | 56.78 (6.02)
  Change: number analyzed (Participants) | 45 | 44
  Change | -3.58 (4.32) | -4.44 (7.07)

12. Secondary Outcome: Change in Healthy Minds Index (HM Index): Awareness
Description: The HM Index assesses qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. There are 4 awareness items. Mean item scores are reported with a range from 0 to 4 where higher scores indicate more awareness.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 3.29 (0.53) | 3.26 (0.67)
  T2 Post-Test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-Test Week 4 | 3.42 (0.66) | 3.40 (0.70)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.13 (0.65) | 0.12 (0.77)

13. Secondary Outcome: Change in Healthy Minds Index (HM Index): Connection
Description: The HM Index assesses qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. There are 6 connection items. Mean item scores are reported with a range from 0 to 4 where higher scores indicate more connection.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 3.56 (0.58) | 3.55 (0.55)
  T2 Post-Test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-Test Week 4 | 3.72 (0.71) | 3.87 (0.44)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.16 (0.48) | 0.34 (0.48)

14. Secondary Outcome: Change in Healthy Minds Index (HM Index): Insight
Description: The HM Index assesses qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. There are 3 insight items. Mean item scores are reported with a range from 0 to 4 where higher scores indicate more insight.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 2.86 (0.68) | 2.77 (0.60)
  T2 Post-Test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-Test Week 4 | 3.11 (0.76) | 3.33 (0.65)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.27 (0.76) | 0.56 (0.80)

15. Secondary Outcome: Change in Healthy Minds Index (HM Index): Purpose
Description: The HM Index assesses qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. There are 4 purpose items. Mean item scores are reported with a range from 0 to 4 where higher scores indicate more purpose.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 3.43 (0.85) | 3.49 (0.83)
  T2 Post-Test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-Test Week 4 | 3.80 (0.79) | 3.88 (0.90)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.38 (0.90) | 0.40 (0.94)

16. Secondary Outcome: Change in Wellbeing Growth Mindset
Description: Well-being Growth Mindset is a 3-item questionnaire assessing participants' perception of the malleability of wellbeing. It is scored on a 1- to 6-point Likert scale where 1 = strongly disagree and 6 = strongly agree. Total scores range from 3 to 18 where higher scores indicate more of a growth mindset (i.e., wellbeing is malleable).
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 13.77 (3.02) | 13.48 (2.99)
  T2 Post-time Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-time Week 4 | 14.60 (2.64) | 15.11 (2.63)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.68 (2.15) | 1.59 (2.38)

17. Secondary Outcome: Change in Five Facet Mindfulness Questionnaire (FFMQ) Awareness Subscale
Description: FFMQ Awareness is a 8-item questionnaire assessing mindful awareness. It is scored on a 1- to 5-point Likert scale where 1 = never or very rarely true and 5 = very often or always true. Mean scores are reported with a range from 1 to 5 where higher scores indicate more mindful awareness.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 3.04 (0.59) | 2.91 (0.91)
  T2 Post-test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-test Week 4 | 3.22 (0.71) | 3.30 (0.74)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.16 (0.63) | 0.37 (0.81)

18. Secondary Outcome: Change in NIH Toolbox Loneliness
Description: NIH Toolbox Loneliness is a 5-item questionnaire assessing loneliness. It is scored on a 1- to 5-point Likert scale where 1 = never and 5 = always. Mean scores are reported for a range from 1 to 5 where higher scores indicate more loneliness.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 2.76 (0.92) | 2.82 (1.01)
  T2 Post-test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-test Week 4 | 2.20 (1.02) | 2.11 (0.87)
  Change: number analyzed (Participants) | 45 | 44
  Change | -0.54 (0.65) | -0.75 (0.99)

19. Secondary Outcome: Change in Experiences Questionnaire (EQ) Decentering Subscale
Description: Experiences Questionnaire Decentering is an 11-item questionnaire assessing the psychological capacity of decentering. It is scored on a 1- to 5-point Likert scale where 1 = never and 5 = all the time. Mean scores are reported for a total range from 1 to 5 where higher scores indicate more decentering.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 2.85 (0.53) | 3.06 (0.55)
  T2 Post-test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-test Week 4 | 3.30 (0.68) | 3.56 (0.63)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.46 (0.55) | 0.52 (0.71)

20. Secondary Outcome: Change in Meaning in Life Questionnaire (MLQ) Presence Subscale
Description: MLQ Presence is a 5-item questionnaire assessing the presence of meaning in life. It is scored on a 1- to 7-point Likert scale where 1 = absolutely untrue and 7 = absolutely true. Mean scores are reported for a total range from 1 to 7 where higher scores indicate greater presence of meaning in life.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
score on a scale
  T1 Baseline | 3.58 (147) | 3.62 (1.50)
  T2 Post-test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-test Week 4 | 4.27 (1.36) | 4.53 (1.31)
  Change: number analyzed (Participants) | 45 | 44
  Change | 0.74 (1.08) | 0.93 (1.29)

21. Secondary Outcome: Change in PROMIS Sleep Disturbance
Description: Sleep disturbance will be assessed using the computer adaptive version of the PROMIS Sleep Disturbance measure. This measure produces scores a T-score with a mean of 50 and a standard deviation of 10. Higher scores indicate greater sleep disturbance.
Time Frame: Baseline, and post-test (week 4)
Population: 3 participants withdrew from the study
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 46 | 46
T-score
  T1 Baseline | 55.56 (7.04) | 53.77 (5.81)
  T2 Post-Test Week 4: number analyzed (Participants) | 45 | 44
  T2 Post-Test Week 4 | 50.23 (8.70) | 48.84 (8.19)
  Change: number analyzed (Participants) | 45 | 44
  Change | -5.20 (6.72) | -5.04 (9.31)

22. Secondary Outcome: Count of Participant Responses to Adverse Event Relevant Survey Item
Description: Participants were asked a single survey item to assess their meditation experience. The query was "I had challenging, difficult, or distressing experiences as a result of my meditation during this study." Participants chose from the following responses: Never, Rarely, Occasionally, Regularly, or Frequently. Count of participants in each arm answering each response is reported here.
Time Frame: up to 4 weeks
Population: 3 participants withdrew from the study prior to the post-test measure, 1 participant did not answer the question
Measure: Count of Participants; unit: Participants
Arm/Group | 5-minute App Usage | 15-minute App Usage
Number analyzed (Participants) | 44 | 44
Participants
  Never | 30 | 33
  Rarely | 9 | 5
  Occasionally | 4 | 4
  Regularly | 1 | 1
  Frequently | 0 | 1

23. Other Pre Specified Outcome: Change in EMA-assessed Psychological Distress (Composite of Depression and Anxiety Items)
Description: A single item reflecting depression and a single item reflecting anxiety are scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much.
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Change in EMA-assessed Mindfulness of Activities
Description: A single item mindfulness of activities is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much.
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Change in EMA-assessed Mindfulness of Feelings / Emotions
Description: A single item assessing awareness of feelings is scored on a 1- to 5-point Likert scale where 1 = not at all aware and 5 = extremely aware.
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Change in EMA-assessed Loneliness
Description: A single item assessing loneliness is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much.
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Change in EMA-assessed Connection With Others
Description: A single item assessing connection with others is scored on a 1- to 5-point Likert scale where 1 = not often at all and 5 = extremely often
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Change in EMA-assessed Decentering
Description: A single item assessing decentering (i.e., experiencing thoughts more as events than direct reflection of reality) is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much.
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Change in EMA-assessed Insight
Description: A single item assessing insight is scored on a 1- to 5-point Likert scale where 1 = not at all aware and 5 = extremely aware
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Change in EMA-assessed Purpose
Description: A single item assessing purpose is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Change in EMA-assessed Stressor Exposure
Description: A single item assessing stressor exposure is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much.
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Change in EMA-assessed Personal Values / Meaning
Description: A single item assessing reflection of personal values in current activity is scored on a 1- to 5-point Likert scale where 1 = not at all reflected and 5 = extremely reflected.
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Change in EMA-assessed Rumination
Description: A single item assessing rumination is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Change in EMA-assessed Informal Practice
Description: A single item assessing application of meditation techniques in daily life (informal practice) is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much.
Time Frame: 4 times per day from baseline to post-test (week 4)
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Change in Pre- and Post-practice Positive Affect
Description: Two items assessing positive affect are scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much.
Time Frame: Before and after meditation practices between baseline and post-test (week 4)
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Change in Pre- and Post-practice Negative Affect
Description: Two items assessing negative affect are scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = very much
Time Frame: Before and after meditation practices between baseline and post-test (week 4)
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Change in Post-practice Focus
Description: A single item assessing focus during meditation is scored on a 1- to 7-point Likert scale where 1 = not at all and 7 = most of the time
Time Frame: Before and after meditation practices between baseline and post-test (week 4)
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Digital Working Alliance Inventory (DWAI)
Description: The DWAI is a 6-item questionnaire assessing participants' alliance with the HMP app. It is scored on a 1- to 7-point Likert scale where 1 = strongly disagree and 7 = strongly agree. Total scores range from 6 to 42 where higher scores indicate a stronger working alliance.
Time Frame: Post-test (week 4)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 4 weeks on study
Description: A single survey item was asked of participants "I had challenging, difficult, or distressing experiences as a result of my meditation during this study". Participants could answer Never, Rarely, Occasionally, Regularly, or Frequently. Please see Secondary Outcome Measures for count of participant responses.
Arm/Group | 5-minute App Usage | 15-minute App Usage
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

LIMITATIONS AND CAVEATS:
This study was not powered to detect between-group differences on pre-post outcomes. Here results are reported by arm for descriptive purposes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT05229406/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT05229406/SAP_001.pdf
  • Informed Consent Form (2022-02-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT05229406/ICF_002.pdf